CLINICAL TRIAL: NCT00246610
Title: A Phase IV, Non-Randomized, Open-Label Trial Evaluating The Safety Of 625 mg Formulation Of VIRACEPT When Administered To HIV-Infected Women During Pregnancy
Brief Title: Safety Of VIRACEPT® 625mg Administered To HIV-Infected Women During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4301017
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infection
Keywords: Non-randomized open-label single-arm study of Nelfinavir plus Combivir in pregnant females infected with HIV-1 virus.
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-label (Experimental): Non-randomized, open-label, single-arm
  Interventions: Drug: Nelfinavir mesylate, 625 mg

INTERVENTIONS:
Drug: Nelfinavir mesylate, 625 mg — Nelfinavir 625 mg [dosed orally as 1250 mg BID (two 625 mg tablets given orally BID)] plus Combivir (lamivudine 150 mg plus zidovudine 300 mg BID dosed orally) administered with food. Subjects will start treatment at their baseline visit. Subjects will be treated for up to 26 weeks during pregnancy plus 6 weeks postpartum.
  Other Names: VIRACEPT plus Combivir

SUMMARY:
This study is an evaluation of the safety of 625 mg formulation when administered to HIV-infected pregnant women from their second trimester through six weeks postpartum. The study will also evaluate the pharmacokinetics of VIRACEPT

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Second trimester of pregnancy

Exclusion Criteria:

* Major current or prior history of obstetrical complications
* Serious current medical diseases
* Evidence of HIV virus resistance to antiretroviral agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Presence or absence of at least one adverse event related to or possibly related to nelfinavir of Grade 2 or greater severity as defined by the DAIDS Table for Grading of Severity of Adult Adverse Experiences in the gastrointestinal or hepatic category | 32 Weeks

SECONDARY OUTCOMES:
Development of primary or active site protease and nucleoside reverse transcriptase inhibitor-associated resistance mutations assessed using standard HIV genotype test on maternal plasma samples | 32 Weeks
Presence or absence of at least one adverse event of Grade 3 or 4 severity in the hematologic, cardiovascular or metabolic categories defined by DAIDS Table or in the dermatologic category as defined by the Supplemental Toxicity Table | 32 Weeks
Adverse pregnancy events which cannot be directly attributed to another cause other than study treatment after consultation with Pfizer Clinician and Site Investigator | 32 Weeks
Adherence assessed using the NIAID ACTG Adherence Modules and by returned medication counts | 32 Weeks
12-hour pharmacokinetic evaluation of nelfinavir | 32 Weeks
Maternal plasma HIV RNA | 32 Weeks
Immunologic response as measured by CD4 and CD8 cell count | 32 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (5):
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
- Pfizer Investigational Site, Toronto, Ontario, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4301017&StudyName=Safety%20Of%20VIRACEPT%3B%20625%20mg%20Administered%20To%20HIV-Infected%20Women%20During%20Pregnancy